CLINICAL TRIAL: NCT00065923
Title: Topiramate Effects on SIB in Prader-Willi Syndrome
Brief Title: Treatment of Self-Injurious Behavior in Individuals With Prader-Willi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R03HD042818 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2010-08

CONDITIONS: Prader-Willi Syndrome; Self-Injurious Behavior
Keywords: Prader-Willi Syndrome; Self-Injurious Behavior
MeSH Terms: conditions — Prader-Willi Syndrome; Self-Injurious Behavior | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
Prader-Willi syndrome (PWS) is a genetic disorder usually caused by the deletion of a specific gene. One of the symptoms of PWS is self-injurious behavior (SIB); a common form of SIB in PWS patients is skin picking. The injury may be severe enough to require frequent medical attention. This trial will evaluate SIB in individuals with PWS and will test the effectiveness of the drug topiramate to control SIB.

DETAILED DESCRIPTION:
PWS is a neurogenetic disorder resulting from a loss of the paternal-only expressed genes on chromosome 15 (15 q11-13). PWS is characterized by a persistent pattern of SIB, most notably skin picking, that results in frequent medical care and attention. SIB in mental retardation and related developmental disabilities is often monitored by behavioral observation methods. Direct evaluation of skin lesions has been reported to help systematically follow wounds and wound healing. However, there are differences between the type and body location of SIB in individuals with PWS as compared to those with mental retardation. The goal of this study is to characterize SIB in PWS and to evaluate the efficacy of topiramate versus placebo in attenuating SIB in individuals with PWS.

A preliminary 8-week open-label study conducted to evaluate topiramate for appetite and weight in PWS has shown good tolerability and beneficial effects of topiramate. During that study, an unexpected and serendipitous finding was that of the six participants, four engaged in SIB and all four had noticeable symptom improvement during the 8 weeks of treatment. Three of these four have continued on topiramate therapy long term with positive results in terms of decreased self-injury.

Participants in the study will be randomized to receive either topiramate or a placebo for 6 weeks. All participants will be monitored for SIB by observation and photographic recordings of the resultant skin lesions, by reports of group home staff, and by standardized rating measurements of self-injury. At the end of 6 weeks, participants receiving topiramate will receive decreasing doses of topiramate; participants receiving placebo will continue to receive the placebo. At week 9, participants previously receiving topiramate will be given placebo and participants previously receiving placebo will be given topiramate. After 6 weeks, all participants will be entered into a 4-month open-label extension phase. Safety and efficacy measurements will be assessed during the 15 study visits; in the event of worsening SIB, the blind will be broken by the study's medical oversight physician and, if appropriate, the participant will be placed directly into the 4-month open-label extension phase.

ELIGIBILITY:
Inclusion Criteria

* PWS due to deletion of 15 q11-13 or uniparental disomy
* Actively engaging skin picking behavior
* Individual with PWS or legal guardian able to provide full informed consent. If legal guardian gives informed consent, then individual with PWS will give his/her assent.
* Acceptable methods of contraception

Exclusion Criteria

* Pregnant or breastfeeding
* Clinically significant suicidality or homicidality
* DSM-IV diagnosis of substance abuse or dependence within 6 months of study entry
* Cardiovascular, hepatic, renal, gastrointestinal, pulmonary, metabolic, endocrine, or other systemic disease which could interfere with treatment or assessment of PWS
* Treatment with any drug which might interact adversely with topiramate
* Medication or significant behavioral management change within 4 weeks of study entry
* Personal history or a first-degree family history of nephrolithiasis

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2002-07; Primary Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan A. Shapira, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida-Brain Institute, Gainesville, Florida, United States

REFERENCES:
- See also: Primary family support organization for Prader-Willi Syndrome — http://www.pwsausa.org